CLINICAL TRIAL: NCT06614881
Title: Optimal Effective Dose of Dexmedetomidine on Postoperative Delirium and Cognitive Function of Elderly Patients Planned For TKA Surgery
Brief Title: Dexmedetomidine Dosage for Postoperative Delirium and Cognitive Function in Elderly TKA Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed B. Abo elkheer, Lecturer of Anesthesiology, Pain, and ICU Department, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36264PR790/7/24
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Post Operative Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (Placebo Comparator)
  Interventions: Drug: Normal saline
- Group D-1 (Active Comparator)
  Interventions: Drug: Dexmedetomidine Injection [Precedex]; Drug: Dexmedetomidine in 0.9 % NaCl 1,000 Mcg/250 mL (4 Mcg/mL) INTRAVEN INFUSION BOTTLE (ML)
- Group D-2 (Active Comparator)
  Interventions: Drug: Dexmedetomidine Injection [Precedex]; Drug: Dexmedetomidine in 0.9 % NaCl 1,000 Mcg/250 mL (4 Mcg/mL) INTRAVEN INFUSION BOTTLE (ML)
- Group D-3 (Active Comparator)
  Interventions: Drug: Dexmedetomidine Injection [Precedex]; Drug: Dexmedetomidine in 0.9 % NaCl 1,000 Mcg/250 mL (4 Mcg/mL) INTRAVEN INFUSION BOTTLE (ML)

INTERVENTIONS:
Drug: Dexmedetomidine Injection [Precedex] — Dexmedetomidine (Precedex, 100 µg/ml) was provided as an intravenous (IV) loading dose of 1 µg/kg over 10-min
  Arms: Group D-1; Group D-2; Group D-3
Drug: Dexmedetomidine in 0.9 % NaCl 1,000 Mcg/250 mL (4 Mcg/mL) INTRAVEN INFUSION BOTTLE (ML) — Dexmedetomidine infusions were prepared to provide 0.5 µg/kg/h
  Arms: Group D-1
Drug: Dexmedetomidine in 0.9 % NaCl 1,000 Mcg/250 mL (4 Mcg/mL) INTRAVEN INFUSION BOTTLE (ML) — Dexmedetomidine infusions were prepared to provide 0.7 µg/kg/h
  Arms: Group D-2
Drug: Dexmedetomidine in 0.9 % NaCl 1,000 Mcg/250 mL (4 Mcg/mL) INTRAVEN INFUSION BOTTLE (ML) — Dexmedetomidine infusions were prepared to provide 1.1 µg/kg/h
  Arms: Group D-3
Drug: Normal saline — loading dose of saline was injected 10-min before induction of anesthesia.
  Arms: Control Group

SUMMARY:
This study aims to evaluate the efficacy of dexmedetomidine in reducing the incidence of postoperative delirium and cognitive dysfunction in elderly patients undergoing total knee arthroplasty (TKA). The study will compare the outcomes of patients receiving dexmedetomidine to those receiving a standard anesthetic or sedative, focusing on factors such as patient characteristics, surgical duration, and postoperative care. The research will explore the potential neuroprotective effects of dexmedetomidine and its ability to mitigate the risks associated with anesthesia and surgery in vulnerable elderly populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Severe chronic knee osteoarthritis inducing limitation of movement and required knee replacements;
* Patients of American Society of Anesthesiologists Classification grades II-III;
* Patients free of exclusion criteria.

Exclusion Criteria:

* Patients of American Society of Anesthesiologists Classification grade >III;
* Patients show a high risk for getting Post Operative Delirium or have severe cognitive dysfunction;
* Patients had a history of uncompensated cardiac, renal, or hepatic diseases;
* Patients had uncontrolled diabetes mellitus or hypertension;
* Patients had other causes for limited movement;
* Patients had autoimmune disease, coagulopathy, severe anemia with a hemoglobin concentration of <7 g%;
* Patients had local bone disorders that may prevent prosthesis stability;
* Patients had allergies or contraindications to the study drugs.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reporting at least a 50% reduction of Postoperative Delirium (measured by Confusion Assessment Method, Delirium Index) post-Total knee arthroplasty under sevoflurane inhalational anesthesia. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El Gharbyia, Egypt